CLINICAL TRIAL: NCT01623453
Title: A Follow-up Study to Evaluate the Sustained Healing Effect the Patients Who Showed Complete Closure of Fistula the Previous ANTG-ASC-210 Study
Brief Title: Follow-up Study of Autologous Adipose-derived Stem Cells (ANTG-ASC) for the Complex Fistula (ANTG-ASC-211)
Acronym: ANTG
Status: Terminated | Type: Observational
Why Stopped: Difficulty recruiting subjects
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ANTG-ASC-211
Record Dates: First submitted 2012-06-08; First posted 2012-06-20 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2012-06

CONDITIONS: Perianal Fistula; Primary; Complex
Keywords: crohn's disease; fistula; complex
MeSH Terms: conditions — Crohn Disease; Fistula | interventions — Population Groups

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Low dose group: Group1. Low dose group
  Interventions: Biological: Autologous adipose derived stem cells(low dose group)
- High dose group: Group2. High dose group
  Interventions: Biological: Autologous adipose derived stem cells(high dose group)

INTERVENTIONS:
Biological: Autologous adipose derived stem cells(low dose group) — low dose group: 1x10e7 cells/mL At 6 weeks after first stem cell injection, fistula closing was assessed. If it is not completely closed, second injection would be applied in 2 weeks. Additional dosage would be doubled to first dosage.
  Other Names: mesenchymal stem cell, ANTG-ASC, adipose derived stem cell; Group 1: low dose group
  Groups: Low dose group
Biological: Autologous adipose derived stem cells(high dose group) — high dose group: 2x10e7 cells/mL At 6 weeks after first stem cell injection, fistula closing was assessed. If it is not completely closed, second injection would be applied in 2 weeks. Additional dosage would be doubled to first dosage.
  Other Names: mesenchymal stem cell, ANTG-ASC, adipose derived stem cell; Group 2: high dose group
  Groups: High dose group

SUMMARY:
This is an open follow-up clinical trial to evaluate a sustained efficacy and safety of ANTG-ASC injection for 4 months (6 months after final dose injection) after Phase II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* the patients who have participated in ANTG-ASC-210 clinical trial
* the patients with complete closure at week 8 after last injection in ANTG-ASC-210 trials
* the patients who submit written informed consents and is able to obey requirements of trials

Exclusion Criteria:

* a patient who has a history of variant Creutzfeldt Jacobs disease or related diseases
* a patient who is allergic to anesthetics, bovine derived proteins or a fibrin glue
* a patient who has an autoimmune disease
* a patient who has infectious diseases such as hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV)
* a patient who has a symptom of septicemia or active tuberculosis (contain tuberculosis of anus and rectum)
* a patient who is pregnant or breast feeding
* a patient who is not willing to use effective contraceptive methods during the study
* a patient who has inflammatory Bowel disease
* a patient who is sensitive to fibrin glue
* a patient who have a clinically relevant history of abuse of alcohol or drugs, habitual smoker (who smoked more than 20 cigarettes a day)
* a patient who is not able to understand the objective of this study or to comply with the study requirements
* a patient who is considered to have a significant disease which can impact the study by investigator
* a patient who is considered not suitable for the study by investigator
* a patient who had a history of surgery for malignant tumor within the last five years (except carcinoma in situ)
* a patient who has multisystemic wasting syndrome (such as tuberculosis, Diabetes, Thyroid disorders, tumor, etc.)
* a patient who has taken cytotoxic drugs (such as immunosuppressants, corticosteroid, cytotoxic chemotherapy, anticoagulants, etc.) during long-term

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: • the patients with complete closure at week 8 after last injection in ANTG-ASC-210 trials
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with Sustained efficacy of complete closure of fistula | Month 4
  Proportion of patients with completely closed of fistula (Month 4)

SECONDARY OUTCOMES:
Number of patients with sustained efficacy of closure of fistula | Month 2, 4
  Proportion of patients with completely closed of fistula (Month 2)
  Proportion of patients with more than 50% closed of fistula (Month 2, 4)
Evaluation of Fecal Incontinence Score | Month 4
  Evaluation of Fecal Incontinence Score (Wexner Score, Cleveland Clinic Continence Scoring System)
Grade of Investigator's satisfaction | Month 2, 4
  Grade of Investigator's satisfaction (Month 2, 4)
  1. very satisfied
  2. satisfied
  3. moderately satisfied
  4. dissatisfied
  5. very dissatisfied
Number of patients with adverse events as a measure of systemic tolerance and physical examinations | Month 2, 4
  1. systemic tolerance (Month 4) (Biochemistry: Albumin, Alkaline phosphatase, ALT, AST, Bilirubin, Calcium, Chloride, Bicarbonate, Creatinine, Glucose, LDH, Potassium, Sodium, Total protein, Urea nitrogen(BUN), Uric acid / Hematology: Hemoglobin, Hematocrit, Reticulocyte count, complete blood cell count with differential, platelet count, WBC with differential count, ESR, PT/APTT)
  2. Physical examination
  3. Pregnancy testing (Month 4)

CONTACTS AND LOCATIONS:
Overall Officials: KJ Park, Principal Investigator — Seoul National University Hospital; DS Kim, Principal Investigator — Daehang Hospital
Locations (2):
- South Korea (2):
  - DaeHang Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided